CLINICAL TRIAL: NCT05354739
Title: A Randomized Clinical Trail Comparing the Effect of Vibration Cold (BUZZY) Device With EMLA Cream in Decreasing the Needle-Related Pain and Anxiety in Pediatric Emergency Setting: a Non-inferiority Study.
Brief Title: Comparing Buzzy Device With Emla Cream in Needle Related Pain
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-20-053
Record Dates: First submitted 2022-04-12; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-02

CONDITIONS: Procedural Pain
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emla Group: Emla Cream
  1 gm of EMLA cream contains lidocaine 25 mg, prilocaine 25 mg, and macrogol glycerol hydroxy stearate. Act as a surface anesthetic of the skin. Will apply ½ tube (approximately 2 gram) per 10 square cm and covered with occlusive dressing. Applied for 30-45 minutes for children needing IV catheter placement or blood extraction based on the treating physician decision depending on the patient's need
  Interventions: Device: The vibration cold device (BUZZY)
- Buzzy Device Group: Buzzy Device
  The vibration cold device (BUZZY) is 8.4 cm X 5.3 cm X 2.9 cm dimensions, exist in different but the investigators will choose the most attractive color, and can be handled by the child prior the procedure
  It composed of two parts:
  * The main body which can be operated by a switch. It generates vibration using two AAA batteries.
  * Removable ice wings. The ice wings are reusable for about 100 times, both wings weighing 18 grams. It stays frozen at room temperature for around 10 minutes. The research nurse will follow the manufactures recommendations (MMJ labs, Atlanta, Georgia, USA).
  Interventions: Device: The vibration cold device (BUZZY)

INTERVENTIONS:
Device: The vibration cold device (BUZZY) — If the patient fulfils the inclusions criteria, the research nurse will obtain informed consent from a parent or legal guardian and assent form if the child is 7years or older. She will assess the ability of the child to use the Faces Pain Scale-Revised (FPS-R), as a pain assessment instrument used by the child. It is a six cartoon faces showing a normal facial expression if no pain, progressing into the facial expression with very severe pain. FPS-R is graded from zero to ten; the child will be asked to quantify the pain by: no hurt, hurt, or very much hurt. This scale is widely used not only in research but also in a routine bases in ours and other units by the nursing staff and are familiar with it. The research nurse is one of the nurses used the same scale during the routine work and will be trained further to ensure consistency, she will document the findings prior, during and after the procedure. This instrument was reliable, valid, and standardized

SUMMARY:
This randomized controlled study will enroll the eligible patients to either the Buzzy device arm or to the EMLA cream arm as a standard therapy. This will be done with concealment; however, blinding will not be practical. Will include 300 participants with 150 in each arm in Al Saad pediatric emergency. The research nurse will use a known valid and reliable measurements scales for the pain and anxiety. The data will be recorded with timing in a prepared form, The SPSS 22.0 and Epi-info soft wares and appropriate statistical tests will be used and will consider P value of <0.05 is statistically significant. The investigators are anticipating a Buzzy device effectiveness to be not less than the EMLA cream but the rapidity of effectiveness in buzzy device of around one minute compared to 30-45 minutes of EMLA cream will be an important outcome in a busy emergency department.

DETAILED DESCRIPTION:
Currently there is strong evidence that children regardless the age feel pain. Research were done and still going on to handle the barriers for pain management in children. Several pain management tools were established but with limitation in efficacy or practicality. EMLA cream, is a mixture of lidocaine and procaine, currently used for pain relief due to needle-related procedures but it needs minimum 30-45 minutes to work. Buzzy is a device that generate vibration with cold leading to pain relief in based on known theories and effective in a minute.

This is non-inferiority study will compare the Buzzy device effectiveness with the EMLA cream, comparing the degree of the child anxiety at different stages of the procedure, and other secondary outcomes. Children 2-14 years of age in need for blood extraction or intravenous cannula insertion, based on their clinical needs, will be included. Determined exclusion criteria will be applied. This randomized controlled study will enroll the eligible patients to either the Buzzy device arm or to the EMLA cream arm as a standard therapy. This will be done with concealment; however, blinding will not be practical. Will include 300 participants with 150 in each arm in Al Saad pediatric emergency. The research nurse will use a known valid and reliable measurements scales for the pain and anxiety. The data will be recorded with timing in a prepared form, The SPSS 22.0 and Epi-info soft wares and appropriate statistical tests will be used and will consider P value of <0.05 is statistically significant. The investigators are anticipating a Buzzy device effectiveness to be not less than the EMLA cream but the rapidity of effectiveness in buzzy device of around one minute compared to 30-45 minutes of EMLA cream will be an important outcome in a busy emergency department

ELIGIBILITY:
Inclusion Criteria:

* All children attending Al Saad PEC with age of 2 up to 14 years of age. Decision made by the treating physician in the PEC for IV catheter placement or blood extraction

Exclusion Criteria:

* Older than 14 years of age or younger than 2 years of age.

  * Children who require immediate emergency intervention, category 1 and 2 in the Canadian Triage and Acuity Scale.
  * Diseases rendering patient to be sensitive to cold such as Sickle Cell disease or patients with Reynaud's phenomena.
  * Skin damage of any degree in the limb where the needle will be inserted.
  * Patients with abnormal sensation in the targeted limb for needle insertion.
  * Any degree of neurological, psychological, or psychiatric disability.
  * Received simple analgesics, paracetamol and nonsteroidal anti-inflammatory drugs within 6 hours prior the procedure.
  * Received procedural sedation/analgesia, any sedative, opioid analgesic, or dissociative drug such as ketamine within 4 hours from the needle prick. Known hyper sensitivity to local anesthetics or any conditions that need precautions to EMLA cream such as G-6PD deficiency, methemoglobinemia, atopic dermatitis or other skin lesion in the needle prick site, patient using antiarrhythmic drug such as amiodarone.
  * Refusal of signing the consent.Known hyper sensitivity to local anesthetics or any conditions that need precautions

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be conducted in Al Saad Pediatric Emergency center (PEC) for all children between the age group of 2 to 14 years.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
To find the difference in needle related pain reduction between Buzzy Device and Emla cream using FLACC pain scale | 1 year
  The Face, Legs, Activity, Crying, Consolability (FLACC) scale is used as an observational scale for pain assessment by the research nurse and a parent. It composed of five behaviors, each is assessed by scoring 0 to 10, based on the pain severity
To find the difference in anxiety reduction by using Observational Scale of Behavioral Distress (OSBD). | 1 year
  Distress scores were calculated by summing the number of 15-second intervals during which each distress behavior occurred and multiplying that number by an expert-determined intensity weight from 1 to 4 reflecting the severity of the behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Haidar, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- [Derived] Haidar NA, Al Amri MH, Sendad NG, Toaimah FHS. Efficacy of Buzzy Device Versus EMLA Cream for Reducing Pain During Needle-Related Procedures in Children: A Randomized Controlled Trial. Pediatr Emerg Care. 2024 Mar 1;40(3):180-186. doi: 10.1097/PEC.0000000000002965. Epub 2023 May 11. PMID 37163686